CLINICAL TRIAL: NCT02407470
Title: A Multicenter, Randomized, Controlled Study of the Efficacy and Safety of the Combination of Adipose Tissue-derived Hematopoietic Stem Cells (AD-HSCs) and ATG in the Treatment of Severe Aplastic Anemia
Brief Title: Safety and Efficacy of Patient's Own AD-MSC and AD-HSC Transplantation in Patients With Severe Aplastic Anemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Collaborators: Peking Union Medical College Hospital (Other); General Hospital of Beijing PLA Military Region (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Qinwei Yin, Professor, General Hospital of Beijing PLA Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ginkgocell-ADHSC-AA-001
Record Dates: First submitted 2015-03-25; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Severe Aplastic Anemia
Keywords: Severe Aplastic Anemia (SAA), Hematopoietic Stem Cells, HSC Transplantation; ATG, Mesenchymal Stem Cells, Transdifferentiation,
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rabbit antithymoglobulin （ATG） (Active Comparator): Patient in this arm will receive rabbit ATG at 3.5 mg/kg/dose IV from day -6 to -2 with the goals of ablating host repressive T cells.
  Interventions: Drug: Rabbit antithymoglobulin (ATG)
- Rabbit ATG & AD-MSCs (Experimental): Patient in this arm will receive rabbit ATG at 3.5 mg/kg/dose IV from day -6 to -2 and then patient's own adipose derived mesenchymal stem cells (AD-MSCs) at a dose of 3000000/kg/d on day 1 to 3.
  Interventions: Drug: Rabbit antithymoglobulin (ATG); Procedure: Adipose derived mesenchymal stem cells ( AD-MSCs)
- Rabbit ATG & AD-HSCs (Experimental): Patient in this arm will receive rabbit ATG at 3.5 mg/kg/dose IV from day -6 to -2 and then patient's own AD-MSC transdifferentiated HSCs (AD-HSCs) at a dose of 3000000/kg/d from day 1 to 4.
  Interventions: Drug: Rabbit antithymoglobulin (ATG); Procedure: AD-MSC transdifferentiated HSCs (AD-HSCs)

INTERVENTIONS:
Drug: Rabbit antithymoglobulin (ATG) — Rabbit ATG at 3.5 mg/kg/dose IV is given from day -6 to -2.
  Other Names: ATG
Procedure: Adipose derived mesenchymal stem cells ( AD-MSCs) — Participants will receive rabbit ATG at 3.5 mg/kg/dose IV from day -6 to -2, and then patient's own AD-MSCs at a dose of 3000000 cells/kg/d on day 1-3.
  Other Names: AD-MSCs
  Arms: Rabbit ATG & AD-MSCs
Procedure: AD-MSC transdifferentiated HSCs (AD-HSCs) — Participants will receive rabbit anti-thymocyte globulin at 3.5 mg/kg/dose IV from day -6 to -2, and then patient's own AD-HSCs at a dose of 3000000 cells/kg/d from day 1 to 4.
  Other Names: AD-HSCs
  Arms: Rabbit ATG & AD-HSCs

SUMMARY:
RATIONALE: It has been shown that about 30% of patients do not respond to immunosuppressive therapy or experience recurrence, and graft rejection and graft-versus-host-disease (GVHD) decrease event-free survival to 30% to 50% in the alternative donor (matched unrelated, partially matched family member) transplantation. Although an overall and disease free survival of 85% to 100%, can be obtained in allogeneic blood or bone marrow stem cell transplantation using an human leukocyte antigen (HLA) matched sibling donor, only about 25% of patients have such a donor.

PURPOSE: In an attempt to avoid GVHD, reduce earlier infection rate and decrease regimen-related toxicity while maintaining better engraftment, this study is to evaluate the effectiveness and safety of patient's own adipose-derived mesenchymal stem cell (AD-MSC) or AD-MSC transdifferentiated HSC (AD-HSC) transplant after an immunosuppressive regimen in treating patients who have severe aplastic anemia.

The patient will be in the study for one year for observation and active monitoring. After treatment and active monitoring are over, the patient's medical condition will be followed indefinitely. The principle measures of safety and efficacy will be :

1. Patient survival probability at 3 months, 6 months and 1 year.
2. Engraftment at 3 months, 6 months and 1 year
3. Incidence of graft versus host disease (GVHD), incidence of acute and chronic GVHD and Incidence of earlier infection rate as well as other complications within 6 months and 1 years.

DETAILED DESCRIPTION:
Severe aplastic anemia is characterized by severe deficiencies in peripheral-blood platelets, white cells, and red cells. These defects in mature cells occur because aplastic bone marrow contains severely reduced numbers of hematopoietic stem cells. To date, Hematopoietic stem cell (HSC) transplants are routinely used to treat patients with many different diseases, including various cancers and blood disorders, such as aplastic anemia. The main sources of HSCs are bone marrow, cord blood and peripheral blood. However, challenges include obtaining enough functional HSCs to ensure optimal engraftment, and avoiding immune rejection and other complications associated with allogeneic transplantations. Novel abundant sources of clinical-grade HSCs are therefore being sought.

Our novel studies have demonstrated that adipose-derived mesenchymal stem cells (AD-MSCs) can be converted rapidly (in 4 days) into AD-HSCs on a large scale (2X108-9 cluster of differentiation 34（CD34）positive cells) by transfection of small RNAs to the the early region 1A (E1A)-like inhibitor of differentiation 1 (EID1) in the presence of specific cytokines. In vitro, AD-HSCs expanded efficiently and resembled cord-blood HSCs in phenotype, genotype, and colony-forming ability. In a mouse model, primary and secondary transplantation analysis and repopulating assays showed that AD-HSCs homed to the bone marrow, differentiated into functional blood cells, and showed a long-term ability to self-renew. we show that adipose-derived mesenchymal stem cells (AD-MSCs) can be converted into AD-HSCs by transfection of small RNAs to the E1A-like inhibitor of differentiation 1 (EID1) in the presence of specific cytokines. In vitro, AD-HSCs expanded efficiently and resembled cord-blood HSCs in phenotype, genotype, and colony-forming ability. In a mouse model, primary and secondary transplantation analysis and repopulating assays showed that AD-HSCs homed to the bone marrow, differentiated into functional blood cells, and showed a long-term ability to self-renew. In the safety aspect, we saw no evidence of leukemia, teratoma and other cancers in the blood, testes and subcutaneous tissues of transplanted mice. More importantly, our preliminary data have shown that AD-HSCs can reconstitute hematopoietic function in five patients with severe aplastic anemia. Based on these premilitary studies,, we have determined to conduct a further clinical investigation in multiple medical centers. In this study we plan to enroll up to 90 patients, to make a comprehensive assessment for this new treatment regimen and to show it is equal or superior to the current immunosuppressive regimen. Patients will be in the study for one years for treatment and active monitoring. All patients will be followed until death.

ELIGIBILITY:
Inclusion Criteria:

Male or female recipients must have histopathologically confirmed diagnosis of SAA-I without or with more than 6 months after less than one treatment with ATG. Diagnostic Criteria for Server Aplastic Anemia will be based on the definitions set forth by the international Aplastic Anemia Study Group.

At least two of the following:

Absolute neutrophil count ≤ 0.5 X 109/l, Platelet count ≤ 20 X 109 /l, Anemia with corrected reticulocyte count ≤ 1%, and Bone marrow cellularity ≤ 25%, or bone marrow cellularity ≤ 50% with fewer than 30% hematopoietic cell, Hepatic: alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) no greater than 4 times normal, Bilirubin: no greater than 2 mg/dl, Renal: Creatinine clearance at least 50 ml/min, Cardiovascular: Shortening fraction or ejection fraction at least 40% of normal for age by echocardiogram or radionuclide scan.

No clinically significant comorbid illnesses (e.g., myocardial infarction or cerebrovascular accident).

Exclusion Criteria:

Active and uncontrolled infection, Active bleeding, Severe allergic history of ATG, HIV-1 infection, Pregnancy or breastfeeding, Carbon monoxide lung diffusion capacity (DLCO) <40% predicted, SAA-II, Patients with severe psychological disorders, Recipients of other clinical trials.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Engraftment at 42 days post AD-HSC transplantation for patients with severe aplastic anemia. | 42 days posttransplant
  Absolute neutrophil count > 0.5 X 109/l and Platelet count > 20 X 109 /l without infusion of platelet for 7 days.

SECONDARY OUTCOMES:
To estimate the overall survival (OS) at 1 year following AD-HSC transplantation for Patients with Severe Aplastic Anemia | 1 year
  Number of Subjects Alive at 12 months Post Transplant
Relapse | 1 year post transplant
  Return of SAA during the specified post-transplantation period.
Incidence of chronic graft-versus-host disease | 6 months
  Number of patients with chronic graft-versus-host disease by 6 months and 1 year
Evaluation of the occurrence of secondary malignancies | 6 months post transplant
  Occurring of any tumors during the specified post-transplantation period.
Hematology labs | 12 weeks
  Association between AD-HSC transplantation and response in hemoglobin, platelet, total white blood cell count, and absolute neutrophil count to be evaluate by maximal hemoglobin, platelet, total white blood cell count, and absolute neutrophil counts achieved in patients with severe aplastic anemia
Number of participants with adverse events as a measure of safety and tolerability of intravenous AD-HSC infusion in patients with severe aplastic anemia | weekly untill 12 months
  Adverse events like allergic reactions, infectious diseases, organ dysfunction or other related to AD-HSC infusion will be assessed
Transfusional requirements | weekly untill 6 months
  Units of blood or platelets transfused after AD-HSC infusion will be measured and compared to previously.
To assess treatment related mortality | 12 months
  Number of death after transplantation during the specified post-transplantation period.

CONTACTS AND LOCATIONS:
Overall Officials: james Q Yin, M.D.,Ph.D., Principal Investigator — The military general hospital of Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China